CLINICAL TRIAL: NCT01556737
Title: Effect of Two Different Isoflavone Supplement Preparations on Gene-expression in Postmenopausal Women
Acronym: ISOII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lisette de Groot, (Vera van der Velpen), Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: NL37475.081.11; ISO II study (Other: Wageningen University)
Record Dates: First submitted 2012-01-09; First posted 2012-03-16 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Postmenopause
Keywords: isoflavone; supplement; daidzein; genistein; gene expression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement (Experimental)
  Interventions: Dietary Supplement: High daidzein supplement; Dietary Supplement: High genistein supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: High daidzein supplement; Dietary Supplement: High genistein supplement

INTERVENTIONS:
Dietary Supplement: High daidzein supplement — 8 weeks exposure to the supplement, daily 100 mg of isoflavones
  Other Names: Phyto soya forte - Arkpharma
Dietary Supplement: High genistein supplement — 8 weeks exposure to the supplement, daily 100 mg of isoflavones
  Other Names: Mega Soja - Springfield

SUMMARY:
Alleged benefits experienced after the consumption of soy in Asian countries have been attributed to the isoflavone content of soy products. Amongst other benefits, isoflavones are believed to relieve menopausal symptoms and are therefore often consumed in supplement form in Western countries. These supplements contain relatively high amounts of isoflavones and are on the market in different compositions. The question is whether supplements with different compositions exert similar effects or whether the effects differ substantially.

DETAILED DESCRIPTION:
Intervention study with two substudies; each substudy is a double blind placebo controlled crossover intervention study. The first substudy has two groups: 'high daidzein' supplement versus placebo (n=18) and vice versa (n=18); the second substudy also has two groups 'high genistein' versus placebo (n=18) and vice versa (n=18).

ELIGIBILITY:
Inclusion Criteria:

* Female
* 50-70 years
* menstrual cycle absent for more than 1 year

Exclusion Criteria:

* current use of contraceptives containing hormones
* current use of hormone replacement therapy
* regular soy product use (more than once a week)
* regular isoflavone supplement use (more than once a week)
* current use of medication containing sexhormones or sexhormone-triggering compounds
* current use of anti-inflammatory medicines
* use of antibiotics in the past 3 months
* severe heart disease
* diabetes
* thyroid disorders --> use of medicines for thyroid disorders
* removed thyroid gland
* complete ovarectomy
* prior diagnosis of cancer
* alcohol and drug abuse
* current smoker
* BMI >35 kg/m2
* allergy to soy (products)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Gene-expression in PBMCs | after 8 weeks exposure to supplement vs after 8 weeks exposure to placebo
  after placebo vs after treatment measured by microarrays

SECONDARY OUTCOMES:
Isoflavone levels in plasma | before and after 8 weeks exposure to supplement vs before and after 8 weeks exposure to placebo
  after placebo vs after treatment measured by HPLC
Gene - expression in adipose tissue | after 8 weeks exposure to supplement vs after 8 weeks exposure to placebo
  after placebo vs after treatment measured by QPCR
Isoflavone levels in adipose tissue | after 8 weeks exposure to supplement vs after 8 weeks exposure to placebo
  levels after placebo vs levels after treatment measured by HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Pieter van 't Veer, Prof, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] van der Velpen V, Geelen A, Hollman PC, Schouten EG, van 't Veer P, Afman LA. Isoflavone supplement composition and equol producer status affect gene expression in adipose tissue: a double-blind, randomized, placebo-controlled crossover trial in postmenopausal women. Am J Clin Nutr. 2014 Nov;100(5):1269-77. doi: 10.3945/ajcn.114.088484. Epub 2014 Aug 20. PMID 25332325